CLINICAL TRIAL: NCT02687438
Title: The PIO III Study: In-office Placement of a Steroid-Eluting Implant Immediately Following Ethmoid Sinus Surgery
Brief Title: The PIO (Propel In Office) III Study of In-office Placement of a Steroid-Eluting Implant Immediately Following Ethmoid Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ENT and Allergy Associates, LLP (Other)
Collaborators: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIO III
Record Dates: First submitted 2016-01-26; First posted 2016-02-22 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Sinusitis
Keywords: Steroid-eluting implant Mometasone Furoate
MeSH Terms: interventions — Debridement; Therapeutic Irrigation; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Steroid-releasing sinus implant placement following ethmoidectomy in addition to post-op standard of care (i.e. debridement, irrigation, and topical steroids)
  Interventions: Device: Steroid-releasing sinus implant; Other: Post-op standard of care

INTERVENTIONS:
Device: Steroid-releasing sinus implant — PROPEL (Intersect ENT, Menlo Park, CA) containing 370mcg of mometasone furoate designed for gradual release over 30 days
  Other Names: PROPEL
Other: Post-op standard of care — post-op standard of care including debridement, irrigation, and/or topical steroids
  Other Names: debridement, irrigation, topical steroids (e.g. mometasone furoate)

SUMMARY:
Report on the technical feasibility and outcomes of in-office placement of PROPEL or PROPEL mini implants immediately following ethmoid sinus surgery

DETAILED DESCRIPTION:
The PROPEL mometasone furoate-releasing implant (Intersect ENT, Menlo Park, CA) is the first FDA-approved device for reducing the need for post-operative interventions by maintaining patency and delivering steroid medication directly into the ethmoid cavity following surgery. Five recently published clinical trials have demonstrated that the mometasone furoate-releasing implant placed in the hospital operating room or in the office setting produces statistically significant reductions in inflammation, polyp formation, and postoperative adhesions. In addition, the implant has been found to significantly reduce the need for postoperative prescription of oral steroids and to decrease the frequency of postoperative lysis of adhesions. Minimal adverse effects were reported in these trials.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of CRS (Chronic Rhinosinusitis) based on the 2015 Clinical Practice Guideline for Adult Sinusitis [6]
* Prior ESS (Ethmoid Sinus Surgery) including bilateral total ethmoidectomy at least 90 days prior to being considered for this study
* Planned ESS includes bilateral polypectomy
* ESS including bilateral polypectomy has been successfully completed without significant complication that, in the opinion of the investigator, would confound study results, and the patient's anatomy remains amenable to implant placement.
* Bilateral polyposis (minimum grade 2 on each side) originating from the ethmoid sinus region
* Complaints of at least 2 of the 5 hallmark symptoms of chronic sinusitis: nasal obstruction/congestion, post-nasal discharge, thick nasal discharge, facial pain/pressure, or decreased sense of smell.
* Minimum symptom threshold (Nasal Obstruction/Congestion minimum score of 2 on scale from 0 to 3)
* Failed medical therapy within the preceding 12 months

Exclusion Criteria:

* Not able to give consent
* Oral-steroid dependent condition
* Allergy or intolerance to corticosteroids
* Clinical evidence of bacterial sinusitis or invasive fungal sinusitis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
the change from baseline to day 90 in nasal obstruction / congestion score | baseline and 90 days from surgery
  nasal obstruction/congestion scored by patients
the change from baseline to day 90 in bilateral polyp grade | baseline and 90 days from surgery
  clinical investigator assessed and by an independent reviewer based on video-endoscopy review

SECONDARY OUTCOMES:
Ethmoid Sinus Obstruction | Baseline, Day 14, Day 30, Day 90 and Month 6
  100mm Visual Analogue Scale (VAS) assessed by clinical investigators and by an independent reviewer
Bilateral Polyp Grading | Day 14, Day 30, Month 6
  Bilateral polyp grade assessed by clinical investigator and by an independent reviewer based on video-endoscopy review
Adhesion Scarring Score | Baseline, Day 14, Day 30, Day 90 and Month 6
  assessed by clinical investigators and by an independent reviewer
Inflammation Score | Baseline, Day 14, Day 30, Day 90 and Month 6
  100mm Visual Analogue Scale (VAS) assessed by clinical investigators and by an independent reviewer
Coagulum/ Crusting Score | Baseline, Day 14, Day 30, Day 90 and Month 6
  100mm Visual Analogue Scale (VAS) assessed by clinical investigators and by an independent reviewer
Nasal Obstruction/ Congestion Score | Day 14, Day 30, Month 6
  scored by patients
Sino-Nasal Outcome Test (SNOT 22) | Baseline, Day 14, Day 30, Day 90 and Month 6
  scored by patients
Medication Requirements | Month 6 post-surgery versus Month 6 post-baseline
  evaluate the need for medication, assessed by clinical investigators
Patient Preference Questionnaire | Baseline procedure, Day 90
  patient tolerability and satisfaction assessed by clinical investigators
Implant Placement Success Rate | time of surgery
  successful access to, and placement of PROPEL Sinus Implant to the target site

CONTACTS AND LOCATIONS:
Overall Officials: B.Todd Schaeffer, MD, Principal Investigator — ENT and Allergy Associates, LLP
Locations (4):
- United States (4):
  - ENT and Allergy Associates, LLP, Lake Success, New York
  - ENT and Allergy Associates, LLP, New York, New York
  - ENT and Allergy Associates, LLP, Port Jefferson, New York
  - ENT and Allergy Associates, LLP, White Plains, New York

IPD SHARING:
Plan to Share IPD: No